CLINICAL TRIAL: NCT02495545
Title: A Multi-Center, Randomized, Controlled, Trial of Cerebrospinal Fluid Drainage (CSFD) in Acute Spinal Cord Injury
Brief Title: Cerebrospinal Fluid Drainage (CSFD) in Acute Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Collaborators: University of Miami (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHX 14BN084
Record Dates: First submitted 2015-07-08; First posted 2015-07-13 (Estimated); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Spinal Cord Injury
Keywords: spinal cord injury (SCI)
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CSFD with elevation of MAP (Experimental): Subjects will receive CSFD and elevation of MAP. Treatments will be 120 hours (5 days) from time treatment is initiated (time 0), and within 24 hours of time of injury. Initiation of CSFD will occur after decompression (during surgery) with a target ITP of 10 mmHg. MAP elevation (norepinephrine drip; goal 100-110 mmHg) will start during surgery, simultaneously with CSFD. 10 mL of CSF will be collected daily for routine lab testing. Post-surgery subjects will be transferred to an intensive care unit (ICU) for duration of treatment or longer if clinically indicated. Target MAP will be sustained within 100-110 mmHg for 5 days. Norepinephrine drip will be used to maintain MAP goal. Subjects will receive other treatment per standard of care at the participating investigational sites.
  Interventions: Procedure: CSFD and elevation of MAP
- Maintenance of MAP (Active Comparator): Subjects will receive elevation of MAP (norepinephrine drip; goal 85-90 mm Hg). Target MAP will be sustained within 85-90 mmHg in the control group for 5 days. Duration of elevation of MAP treatment will be 120 hours (5 days) from time treatment is (time 0). Subjects will receive the same treatment as the subjects in investigational arm except for the initiation of the CSFD and less aggressive MAP elevation. They will have a drain placed the same way as the experimental subjects. While drain is in place, 10 mL of cerebrospinal fluid will be collected daily for laboratory testing. After that, ITP will be monitored but CSFD will not be initiated. Subjects will receive other treatment per standard of care at participating investigational sites.
  Interventions: Procedure: Maintenance of MAP

INTERVENTIONS:
Procedure: CSFD and elevation of MAP — Lumbar drain placement with CSFD with elevation of MAP
  Arms: CSFD with elevation of MAP
Procedure: Maintenance of MAP — Lumbar drain placement without CSFD and with maintenance of MAP
  Arms: Maintenance of MAP

SUMMARY:
The purpose of this Phase IIB randomized controlled trial is to evaluate the safety and efficacy of CSFD and to provide a preliminary clinical efficacy evaluation of the combination of CSFD and elevation of mean arterial pressure (MAP) in patients with acute spinal cord injury (SCI). The objectives of the trial are to evaluate (i) efficacy of reducing intrathecal pressure (ITP) by CSFD in patients with acute SCI; (ii) preliminary efficacy of combination of CSFD and elevation of MAP compared to elevation of MAP alone in improving neurologic motor outcomes in patients with acute SCI; and, (iii) safety of intensive CSFD in acute SCI patients.

DETAILED DESCRIPTION:
Acute spinal cord injury (SCI) affects 10,000-14,000 persons per year in the United States (Burke, Linden et al. 2001). There are 150,000-300,000 persons living with significant disabilities from SCI at any given time (Bernhard, Gries et al. 2005). The average age of incident cases of SCI is 47 years and about 78% of the cases are males (DeVivo and Chen 2011). Estimates of the lifetime costs to care for someone with a SCI range from $325,000 to $1.35 million and the yearly cost to society reaches $8 billion (Sekhon and Fehlings 2001). With better long term care technologies, these costs are expected to continue to rise. Although there have been significant advances in accessibility for people with disabilities, the goal of medical science is to overcome the physiological barriers imposed by the injury itself and allow these individuals to regain their pre-injury level of neurological function (Rowland, Hawryluk et al. 2008). The injury to the spinal cord occurs in two phases. The first phase is the primary physical damage due to the impact energy of the compressive nature of the injury. The damage can be very complex with shearing of the axons, destruction of the cell bodies and disruption of the microvasculature at the site of injury. The secondary phase of the injury begins soon after the primary injury has occurred and can be influenced by many factors such as hypoxia, hypotension, and the extent of the primary injury. Spinal cord ischemia post-injury causes a significant increase in cell death and more significant neurological disability. Limiting tissue hypoperfusion post-injury can decrease the amount of cell death and axonal damage. Lumbar cerebrospinal fluid drainage (CSFD) together with increased mean arterial blood pressure (MAP) in the immediate post-injury period can reduce spinal cord tissue hypoperfusion. By reducing spinal cord hypoperfusion through elevation of MAP, less cell death and axonal damage will occur, leading to an improvement in neurological function. The feasibility of CSFD as a means for reducing the intrathecal pressure (ITP) in patients with acute SCI has been demonstrated in a small randomized controlled trial by Kwon et al (Kwon, Curt et al. 2009). The limitations were a small sample size, broad inclusion criteria, lack of statistical power calculation and restricted drainage regimen (maximum 10 mL per hour).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years inclusive;
* Diagnosis of acute SCI;
* Injury is less than 24 hours old;
* ISNCSCI Impairment Scale Grade "A," "B" or "C" based upon first ISNCSCI evaluation after arrival to the hospital;
* Neurological level of injury between C4-C8 based upon first ISNCSCI evaluation after arrival to the hospital;
* Women of childbearing potential must have a negative serum β-hCG pregnancy test or a negative urine pregnancy test;
* Patient is willing to participate in the study;
* Informed consent document signed by patient or witnessed informed consent document;
* No contraindications for study treatment(s);
* Able to cooperate in the completion of a standardized neurological examination by ISNCSCI standards (includes patients who are on a ventilator).

Exclusion Criteria:

* Injury arising from penetrating mechanism;
* Significant concomitant head injury defined by a Glasgow Coma Scale (GCS) score < 14 with a clinically significant abnormality on a head CT (head CT required only for patients suspected to have a brain injury at the discretion of the investigator);
* Pre-existing neurologic or mental disorder which would preclude accurate evaluation and follow-up (i.e. Alzheimer's disease, Parkinson's disease, unstable psychiatric disorder with- hallucinations and/or delusions or schizophrenia);
* Prior history of SCI;
* Recent history (less than 1 year) of chemical substance dependency or significant psychosocial disturbance that may impact the outcome or study participation, in the opinion of the investigator;
* Is a prisoner;
* Participation in another clinical trial within the past 30 days;
* Acquired immune deficiency syndrome (AIDS) or AIDS-related complex;
* Active malignancy or history of invasive malignancy within the last five years, with the exception of superficial basal cell carcinoma or squamous cell carcinoma of the skin that has been definitely treated. Patients with carcinoma in situ of the uterine cervix treated definitely more than 1 year prior to enrollment may enter the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-10; Primary Completion 2019-10-25 (Actual); Study Completion 2019-10-25 (Actual)

PRIMARY OUTCOMES:
Change in ITP | 120 hours
  ITP will be measured in both groups every hour for the duration of study treatment for a total of 121 measurements consisting of one pre-treatment measurement (time 0 hours) and 120 measurements during the treatment (time 1-120 hours).
Change in International Standards for Classification of Spinal Cord Injury Motor Score (ISNCSCI, formerly ASIA) | 180 days
  ISNCSCI Motor Score will be obtained at hospital arrival (baseline), 72 hours post-injury, 84 days and 180 days post-treatment. The primary endpoint is difference between the Motor Score at 180 days and baseline.

SECONDARY OUTCOMES:
ISNCSCI Grade | Change in ISNCSCI grade between 180 days and baseline
ISNCSCI Sensory Scores | Change in ISNCSCI Sensory Scores (Light Touch and Pin Prick) between 180 days and baseline
ISNCSCI Upper Extremity Motor Score | Change in ISNCSCI Upper Extremity Motor Score between 180 days and baseline
ISNCSCI Lower Extremity Motor Score | Change in ISNCSCI Lower Extremity Motor Score between 180 days and baseline
Spinal Cord Independence Measure (SCIM) | Spinal Cord Independence Measure (SCIM) at 180 days
Pain level per patient report | Pain Numeric Rating Scale (NRS) at 180 days
  Using a numeric pain rating scale, subjects will indicate level of pain at time measure occurs

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Theodore, MD, Principal Investigator — Barrow Neurological Institute, St. Joseph's Hospital and Medical Center
Locations (3):
- United States (3):
  - University of Alabama School of Medicine Department of Neurosurgery, Birmingham, Alabama
  - Barrow Neurological Institute St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - University of Arizona Department of Surgery Division of Neurosurgery, Tucson, Arizona

REFERENCES:
- [Background] Amar AP, Levy ML. Pathogenesis and pharmacological strategies for mitigating secondary damage in acute spinal cord injury. Neurosurgery. 1999 May;44(5):1027-39; discussion 1039-40. doi: 10.1097/00006123-199905000-00052. PMID 10232536
- [Background] Bernhard M, Gries A, Kremer P, Bottiger BW. Spinal cord injury (SCI)--prehospital management. Resuscitation. 2005 Aug;66(2):127-39. doi: 10.1016/j.resuscitation.2005.03.005. PMID 15950358
- [Background] Brown PD, Davies SL, Speake T, Millar ID. Molecular mechanisms of cerebrospinal fluid production. Neuroscience. 2004;129(4):957-70. doi: 10.1016/j.neuroscience.2004.07.003. PMID 15561411
- [Background] Burke DA, Linden RD, Zhang YP, Maiste AC, Shields CB. Incidence rates and populations at risk for spinal cord injury: A regional study. Spinal Cord. 2001 May;39(5):274-8. doi: 10.1038/sj.sc.3101158. PMID 11438844
- [Background] Casha S, Christie S. A systematic review of intensive cardiopulmonary management after spinal cord injury. J Neurotrauma. 2011 Aug;28(8):1479-95. doi: 10.1089/neu.2009.1156. Epub 2010 Apr 8. PMID 20030558
- [Background] Coselli JS, LeMaire SA, Koksoy C, Schmittling ZC, Curling PE. Cerebrospinal fluid drainage reduces paraplegia after thoracoabdominal aortic aneurysm repair: results of a randomized clinical trial. J Vasc Surg. 2002 Apr;35(4):631-9. doi: 10.1067/mva.2002.122024. PMID 11932655
- [Background] DeVivo MJ, Chen Y. Trends in new injuries, prevalent cases, and aging with spinal cord injury. Arch Phys Med Rehabil. 2011 Mar;92(3):332-8. doi: 10.1016/j.apmr.2010.08.031. PMID 21353817
- [Background] Dohrmann GJ, Wick KM, Bucy PC. Spinal cord blood flow patterns in experimental traumatic paraplegia. J Neurosurg. 1973 Jan;38(1):52-8. doi: 10.3171/jns.1973.38.1.0052. No abstract available. PMID 4682352
- [Background] Fehlings MG, Tator CH, Linden RD. The relationships among the severity of spinal cord injury, motor and somatosensory evoked potentials and spinal cord blood flow. Electroencephalogr Clin Neurophysiol. 1989 Jul-Aug;74(4):241-59. doi: 10.1016/0168-5597(89)90055-5. PMID 2471626
- [Background] Francel PC, Long BA, Malik JM, Tribble C, Jane JA, Kron IL. Limiting ischemic spinal cord injury using a free radical scavenger 21-aminosteroid and/or cerebrospinal fluid drainage. J Neurosurg. 1993 Nov;79(5):742-51. doi: 10.3171/jns.1993.79.5.0742. PMID 8410254
- [Background] Guha A, Tator CH, Rochon J. Spinal cord blood flow and systemic blood pressure after experimental spinal cord injury in rats. Stroke. 1989 Mar;20(3):372-7. doi: 10.1161/01.str.20.3.372. PMID 2922776
- [Background] Hadley MN, Walters BC. Introduction to the Guidelines for the Management of Acute Cervical Spine and Spinal Cord Injuries. Neurosurgery. 2013 Mar;72 Suppl 2:5-16. doi: 10.1227/NEU.0b013e3182773549. No abstract available. PMID 23417174
- [Background] Hadley MN, Walters BC, Grabb PA, Oyesiku NM, Przybylski GJ, Resnick DK, Ryken TC, Mielke DH. Guidelines for the management of acute cervical spine and spinal cord injuries. Clin Neurosurg. 2002;49:407-98. No abstract available. PMID 12506565
- [Background] Hickey R, Albin MS, Bunegin L, Gelineau J. Autoregulation of spinal cord blood flow: is the cord a microcosm of the brain? Stroke. 1986 Nov-Dec;17(6):1183-9. doi: 10.1161/01.str.17.6.1183. PMID 3810718
- [Background] Horn EM, Theodore N, Assina R, Spetzler RF, Sonntag VK, Preul MC. The effects of intrathecal hypotension on tissue perfusion and pathophysiological outcome after acute spinal cord injury. Neurosurg Focus. 2008;25(5):E12. doi: 10.3171/FOC.2008.25.11.E12. PMID 18980472
- [Background] Kindt GW. Autoregulation of spinal cord blood flow. Eur Neurol. 1971-1972;6(1):19-23. doi: 10.1159/000114459. No abstract available. PMID 5005114
- [Background] Kobrine AI, Doyle TF, Martins AN. Autoregulation of spinal cord blood flow. Clin Neurosurg. 1975;22:573-81. doi: 10.1093/neurosurgery/22.cn_suppl_1.573. PMID 810290
- [Background] Kobrine AI, Evans DE, Rizzoli HV. The role of the sympathetic nervous system in spinal cord autoregulation. Acta Neurol Scand Suppl. 1977;64:54-5. No abstract available. PMID 409084
- [Background] Kwon BK, Curt A, Belanger LM, Bernardo A, Chan D, Markez JA, Gorelik S, Slobogean GP, Umedaly H, Giffin M, Nikolakis MA, Street J, Boyd MC, Paquette S, Fisher CG, Dvorak MF. Intrathecal pressure monitoring and cerebrospinal fluid drainage in acute spinal cord injury: a prospective randomized trial. J Neurosurg Spine. 2009 Mar;10(3):181-93. doi: 10.3171/2008.10.SPINE08217. PMID 19320576
- [Background] Martirosyan NL, Feuerstein JS, Theodore N, Cavalcanti DD, Spetzler RF, Preul MC. Blood supply and vascular reactivity of the spinal cord under normal and pathological conditions. J Neurosurg Spine. 2011 Sep;15(3):238-51. doi: 10.3171/2011.4.SPINE10543. Epub 2011 Jun 10. PMID 21663407
- [Background] Mokri B. The Monro-Kellie hypothesis: applications in CSF volume depletion. Neurology. 2001 Jun 26;56(12):1746-8. doi: 10.1212/wnl.56.12.1746. PMID 11425944
- [Background] Palesch YY, Tilley BC, Sackett DL, Johnston KC, Woolson R. Applying a phase II futility study design to therapeutic stroke trials. Stroke. 2005 Nov;36(11):2410-4. doi: 10.1161/01.STR.0000185718.26377.07. Epub 2005 Oct 13. PMID 16224086
- [Background] Piano G, Gewertz BL. Mechanism of increased cerebrospinal fluid pressure with thoracic aortic occlusion. J Vasc Surg. 1990 May;11(5):695-701. doi: 10.1067/mva.1990.19358. PMID 2335835
- [Background] Ploumis A, Yadlapalli N, Fehlings MG, Kwon BK, Vaccaro AR. A systematic review of the evidence supporting a role for vasopressor support in acute SCI. Spinal Cord. 2010 May;48(5):356-62. doi: 10.1038/sc.2009.150. Epub 2009 Nov 24. PMID 19935758
- [Background] Rowland JW, Hawryluk GW, Kwon B, Fehlings MG. Current status of acute spinal cord injury pathophysiology and emerging therapies: promise on the horizon. Neurosurg Focus. 2008;25(5):E2. doi: 10.3171/FOC.2008.25.11.E2. PMID 18980476
- [Background] Royston P, Barthel FM, Parmar MK, Choodari-Oskooei B, Isham V. Designs for clinical trials with time-to-event outcomes based on stopping guidelines for lack of benefit. Trials. 2011 Mar 18;12:81. doi: 10.1186/1745-6215-12-81. PMID 21418571
- [Background] Ryken TC, Hurlbert RJ, Hadley MN, Aarabi B, Dhall SS, Gelb DE, Rozzelle CJ, Theodore N, Walters BC. The acute cardiopulmonary management of patients with cervical spinal cord injuries. Neurosurgery. 2013 Mar;72 Suppl 2:84-92. doi: 10.1227/NEU.0b013e318276ee16. No abstract available. PMID 23417181
- [Background] Sekhon LH, Fehlings MG. Epidemiology, demographics, and pathophysiology of acute spinal cord injury. Spine (Phila Pa 1976). 2001 Dec 15;26(24 Suppl):S2-12. doi: 10.1097/00007632-200112151-00002. PMID 11805601
- [Background] Senter HJ, Venes JL. Loss of autoregulation and posttraumatic ischemia following experimental spinal cord trauma. J Neurosurg. 1979 Feb;50(2):198-206. doi: 10.3171/jns.1979.50.2.0198. PMID 430132
- [Background] Smith AJ, McCreery DB, Bloedel JR, Chou SN. Hyperemia, CO2 responsiveness, and autoregulation in the white matter following experimental spinal cord injury. J Neurosurg. 1978 Feb;48(2):239-51. doi: 10.3171/jns.1978.48.2.0239. PMID 624973
- [Background] Svensson LG, Crawford ES, Hess KR, Coselli JS, Safi HJ. Experience with 1509 patients undergoing thoracoabdominal aortic operations. J Vasc Surg. 1993 Feb;17(2):357-68; discussion 368-70. PMID 8433431
- [Background] Sydes MR, Parmar MK, Mason MD, Clarke NW, Amos C, Anderson J, de Bono J, Dearnaley DP, Dwyer J, Green C, Jovic G, Ritchie AW, Russell JM, Sanders K, Thalmann G, James ND. Flexible trial design in practice - stopping arms for lack-of-benefit and adding research arms mid-trial in STAMPEDE: a multi-arm multi-stage randomized controlled trial. Trials. 2012 Sep 15;13:168. doi: 10.1186/1745-6215-13-168. PMID 22978443
- [Background] Tator CH. Spine-spinal cord relationships in spinal cord trauma. Clin Neurosurg. 1983;30:479-94. doi: 10.1093/neurosurgery/30.cn_suppl_1.479. No abstract available. PMID 6667588
- [Background] Tator CH, Fehlings MG. Review of the secondary injury theory of acute spinal cord trauma with emphasis on vascular mechanisms. J Neurosurg. 1991 Jul;75(1):15-26. doi: 10.3171/jns.1991.75.1.0015. PMID 2045903
- [Background] Walters BC. Methodology of the Guidelines for the Management of Acute Cervical Spine and Spinal Cord Injuries. Neurosurgery. 2013 Mar;72 Suppl 2:17-21. doi: 10.1227/NEU.0b013e318276ed9a. No abstract available. PMID 23417175
- [Background] Walters BC, Hadley MN, Hurlbert RJ, Aarabi B, Dhall SS, Gelb DE, Harrigan MR, Rozelle CJ, Ryken TC, Theodore N; American Association of Neurological Surgeons; Congress of Neurological Surgeons. Guidelines for the management of acute cervical spine and spinal cord injuries: 2013 update. Neurosurgery. 2013 Aug;60(CN_suppl_1):82-91. doi: 10.1227/01.neu.0000430319.32247.7f. No abstract available. PMID 23839357